CLINICAL TRIAL: NCT03228615
Title: Pilot Trial of a Multi-Component Decision Making Intervention in IBD
Brief Title: IBD Shared Decision Making Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Ellen A. Lipstein MD, MPH, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-8792
Record Dates: First submitted 2017-07-12; First posted 2017-07-25 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: shared decision making
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This clinical trial uses prospective repeated measures in a before-after study design. Following enrollment of the usual care group (i.e., 50% recruitment goal has been reached), physicians will be trained to use the intervention. We will then enroll the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making Intervention (Experimental)
  Interventions: Other: SDM Intervention
- Usual Care Group (No Intervention)

INTERVENTIONS:
Other: SDM Intervention — Intervention Component A: letter to activate families; Intervention Component B: in-clinic decision support; Intervention Component C: follow-up phone call
  Arms: Shared Decision Making Intervention

SUMMARY:
The purpose of this clinical trial is to implement a multi-component shared decision making intervention for families of children with IBD. The main objective of this research will be to assess the acceptability, feasibility and clinical and decision outcomes of a multi-component decision support intervention targeted at families of children with IBD who are making decisions about treatment with TNFαi agents.

DETAILED DESCRIPTION:
Research has shown that when making decisions about treatment with anti-tumor necrosis factor-α (TNFαi) agents, parents of children with inflammatory bowel disease (IBD) experience high levels of decisional conflict. This extreme level of conflict is due to the challenge of considering an effective treatment that has potentially serious side-effects. Elevated levels of decisional conflict have been associated with delays in decision making and failures to implement treatment plans. Given that such delays may lead to worse clinical outcomes, there is an urgent need to improve the decision-making process around TNFαi therapy. The use of structured decision support to help inform and guide parents through this challenging decision may improve the decision-making process. Such structure facilitates high-quality decision making by providing balanced, accurate information, helping individuals clarify what is most important to them, and facilitating conversations between families and healthcare providers. Based the investigators' prior research into the TNFαi decision process, the investigators developed a multi-component decision support intervention designed to improve the TNFαi decision process. This intervention will be tested in a controlled pilot trial designed to assess the acceptability and feasibility of a multi-component intervention and to determine the effect size of the multi-component intervention on both clinical and decision outcomes in children and adolescents with IBD and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Clinician anticipates discussing TNFai treatment at clinic visit; parent and patient willing to have visit video-recorded

Exclusion Criteria:

* patient over age 17; prior use of TNFai; unable to read and speak English; clinic visit not conducted in English; previous participation in this study; known major mental illness in parent or adolescent patient; medical instability at scheduled visit; patient's gastroenterologist is a study investigator

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Acceptability of multi-component intervention: OPTION scale | Baseline
  Measures observed shared decision making based on review of the video-recorded visit
Feasibility of multi-component intervention: Receipt of intervention components | 1 month post baseline
  The percentage of participants who receive each individual component (i.e., pre-visit email/letter, in-clinic decision support, follow-up phone call)
Feasibility of multi-component intervention: Length of clinic visit | Baseline
  Measures the length of the clinic visit with in-clinic decision support intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No